CLINICAL TRIAL: NCT07123285
Title: Effect of Photobiomodulation on the Healing of Venous Ulcers in the Lower Limbs
Brief Title: Effect of Photobiomodulation on Healing of Venous Leg Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE88980225
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Venous Disease; Venous Insufficiency (Chronic)(Peripheral); Venous Insufficiency of Leg; Venous Leg Ulcer (VLU); Venous Leg Ulcer; Venous Hypertension Ulcers; Varicose Ulcers; Varicose Ulcer of Lower Limb
Keywords: venous ulcers; varicose ulcers; photobiomodulation; lasers; phototherapy; venous leg ulcer
MeSH Terms: conditions — Venous Insufficiency; Varicose Ulcer | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, controlled, parallel-group clinical trial with two arms: an Experimental Group receiving photobiomodulation therapy (PBM) plus compression therapy, and a Control Group receiving sham PBM plus compression therapy. Participants are allocated in a 1:1 ratio and will not cross over between groups. Each group receives 32 treatment sessions over a 16-week period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, both the participants and the outcome assessors are blinded to the treatment assignments. However, the nurse administering the photobiomodulation therapy is not blinded and knows the group allocation in order to correctly perform the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation plus Compression Therapy (Experimental): Participants in this arm will receive photobiomodulation therapy using a low-level laser device with 4 emitters operating at 660 nm and 808 nm wavelengths. Each emitter delivers 6 Joules of energy at 100 mW power. Treatment sessions are conducted twice weekly (Monday and Wednesday) for 16 weeks, totaling 32 sessions. In addition, standard compression therapy will be applied as per clinical guidelines for venous leg ulcers.
  Interventions: Device: Photobiomodulation plus Compression Therapy
- Compression Therapy plus Sham Photobiomodulation (Sham Comparator): Participants in this arm will receive sham photobiomodulation therapy using the same laser device but without active laser emission (placebo). Treatment sessions are also conducted twice weekly for 16 weeks, totaling 32 sessions. They will also receive standard compression therapy as per clinical guidelines for venous leg ulcers.
  Interventions: Device: Compression Therapy plus Sham Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation plus Compression Therapy — This intervention uses a low-level laser device with 8 emitters, including 4 red emitters at 660 nm and 4 infrared emitters at 808 nm. Each emitter delivers 6 Joules of energy at 100 mW power, with a total power output of 800 mW. Treatment is administered twice weekly over 16 weeks, totaling 32 sessions per participant. The device is used in combination with standard compression therapy for venous leg ulcer management.
  Other Names: Low-Level Laser Therapy; Photobiomodulation; LLLT; Photobiomodulation Therapy with Low-Level Laser
  Arms: Photobiomodulation plus Compression Therapy
Device: Compression Therapy plus Sham Photobiomodulation — This intervention uses a sham photobiomodulation therapy with the same laser device used in the active group but without emission of therapeutic laser light (inactive device). The device appears identical and the treatment sessions are conducted twice weekly over 16 weeks, totaling 32 sessions per participant. Participants also receive standard compression therapy for venous leg ulcer management. This sham procedure is designed to mimic the active treatment without delivering any laser energy, serving as a placebo control.
  Other Names: Placebo Photobiomodulation; Laser Simulation; Placebo Laser Treatment; Inactive Laser Therapy
  Arms: Compression Therapy plus Sham Photobiomodulation

SUMMARY:
This randomized, controlled, double-blind clinical trial will evaluate the efficacy of photobiomodulation (PBM) combined with compression therapy in the healing of venous ulcers (VUs) in the lower limbs. A total of 96 participants will be allocated into two groups: Experimental Group (PBM + compression) and Control Group (sham PBM + compression). Treatments will be administered twice weekly for 16 weeks (32 sessions). The primary outcome will be complete wound healing. Secondary outcomes include changes in ulcer area and volume, pain (VAS), quality of life (SF-36), clinical severity (VCSS), wound quality (Bates-Jensen Scale), infrared thermography, and treatment costs. Data will be analyzed using ANOVA or Kruskal-Wallis, chi-square or Fisher's exact test, and Kaplan-Meier survival analysis, with a significance level of p < 0.05.

DETAILED DESCRIPTION:
Venous ulcers (VUs) represent a significant public health problem, characterized by prolonged duration, high recurrence rates, and economic, social, and quality-of-life impacts on affected patients. Currently, the most commonly used conventional treatment for VUs includes topical agents, pharmacotherapy, and compression therapy. Photobiomodulation (PBM) has been widely utilized in wound healing techniques, accelerating the healing process and improving patients' quality of life. This study aims to evaluate the efficacy of PBM combined with compression therapy (gold standard) in the healing time of VUs in the lower limbs. This will be a prospective, randomized, controlled, double-blind clinical trial. A total of 96 participants with venous ulcers in the lower limbs will be randomized into two groups: the Experimental Group (n=48), which will receive compression therapy combined with PBM (6 J per emitter, 4 emitters at 660 nm and 808 nm, total power of 400 mW, 100 mW per emitter, twice a week), and the Control Group (n=48), which will receive compression therapy and sham PBM. Patients will be treated twice a week (Monday and Wednesday) as per the routine of the wound care room at the Lençóis Paulista Health Unit. The researcher will conduct the treatment in collaboration with a trained and calibrated nurse. Each patient will receive 32 PBM or sham PBM sessions. Outcomes will be assessed weekly by the same researcher over 16 weeks. If positive results are observed, participants will be invited to undergo the experimental group treatment. At the end of the study, the primary outcome will be complete healing, defined as total re-epithelialization of the skin without drainage or the need for dressings (16 weeks). Secondary outcomes will include changes in wound size (area and volume), the rate of ulcer size reduction, adverse effects, and additional evaluations such as wound quality assessed by the Bates-Jensen Scale, pain intensity measured by the Visual Analog Scale (VAS), and quality of life assessed using the SF-36 questionnaire. Additional analyses will include wound temperature measurement using infrared thermography, clinical changes assessed by the Venous Clinical Severity Score (VCSS), and treatment costs. For objective wound size analysis, the Tissue Analytics® application will be used, enabling automatic measurements through digital images captured via smartphones. Data will be analyzed after assessing normality using either a two-way ANOVA or the Kruskal-Wallis test. Categorical variables will be compared using the chi-square test or Fisher's exact test. Survival analysis for the primary outcome will be conducted using the Kaplan-Meier method and the log-rank test. A significance level of p < 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes;
* Individuals with venous ulcers in the lower limbs for at least three weeks that have not healed;
* Age between 18 and 85 years;
* Residents of Lençóis Paulista or nearby regions.

Exclusion Criteria:

* Patients with ulcers of non-venous etiology;
* Pregnant women;
* Presence of severe arterial disease in the lower limbs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Complete healing or reduction in venous ulcer size | From enrollment to the end of the 16-week treatment period
  Defined as total re-epithelialization of the wound with no drainage and no need for dressings, or a significant reduction in wound size by the end of the treatment period.

SECONDARY OUTCOMES:
Adverse events | From the first treatment session to the end of the 16-week treatment period
  Adverse events will be recorded and classified according to severity (mild, moderate, severe) and relationship to the intervention. Frequency and type of events will be analyzed for both groups.
Wound quality assessment using the Bates-Jensen Wound Assessment Tool | At baseline, week 4, week 8, and week 16
  Wound quality will be assessed using the Bates-Jensen Wound Assessment Tool, which evaluates parameters such as wound size, depth, edges, exudate, and tissue type. Assessments will be conducted at four time points to monitor healing progression.
Pain intensity measured by Visual Analog Scale | Twice per week, over 16 weeks
  Pain intensity will be measured using the Visual Analog Scale (VAS). The VAS is a 10-centimeter line anchored by two extremes: 0 = "no pain" and 10 = "worst imaginable pain." Higher scores indicate greater pain intensity (worse outcome). Measurements will be recorded before and after each laser or sham session. In addition, the frequency and total dosage of paracetamol (acetaminophen) use will be documented throughout the study period to evaluate analgesic consumption related to pain control.
Quality of life assessment using SF-36 questionnaire | At baseline and after 16 weeks
  Quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36), which evaluates eight health domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality, emotional well-being, social functioning, pain, and general health perceptions. Each domain score ranges from 0 to 100, with higher scores indicating better health status and quality of life.
Venous Clinical Severity Score (VCSS) | At baseline, week 4, week 8, and week 16
  Venous disease severity will be assessed using the Venous Clinical Severity Score (VCSS). The VCSS includes 10 clinical domains: pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulcers, size of active ulcers, and use of compression therapy. Each domain is scored from 0 (absent/normal) to 3 (severe), resulting in a total score ranging from 0 to 30. Higher scores indicate greater venous disease severity (worse outcome).
Wound area measurement using ImitoWound® | At baseline, week 4, week 8, and week 16
  Ulcer area will be measured via digital photographs analyzed with the Tissue ImitoWound® mobile application, which automatically calculates wound area through image recognition and calibration.
Total treatment cost | Cumulative from the start of treatment to the end of the 16-week treatment period
  Direct treatment costs will be calculated by totaling the resources used per patient, including laser equipment use, compression therapy, dressings, debridement, and clinical supplies. Cost-effectiveness analysis will be performed between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Ratto Tempestini Horliana, PhD, Study Director — University of Nove de Julho
Locations (1):
- Estratégia da Saúde da Família Monte Azul - "Antonio Benedetti"., Lençóis Paulista, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
I will analyze any request for access to individual participant data and will decide later whether to share it, following ethical guidelines and data privacy regulations.
Supporting Information: Study Protocol
Time Frame: When we have published the data